CLINICAL TRIAL: NCT05791006
Title: Neuropsychology of Financial Capacity
Acronym: NEUROFIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 25C121
Record Dates: First submitted 2023-03-05; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Parkinson Disease; Brain Tumor; Stroke
MeSH Terms: conditions — Parkinson Disease; Brain Neoplasms; Stroke | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients with Parkinson's Disease/Parkinsonisms
  Interventions: Behavioral: Neuropsychological tests
- Patients with brain tumors
  Interventions: Behavioral: Neuropsychological tests
- Patients with ischemic or haemorrhagic stroke
  Interventions: Behavioral: Neuropsychological tests
- Healthy Controls
  Interventions: Behavioral: Neuropsychological tests

INTERVENTIONS:
Behavioral: Neuropsychological tests — Neuropsychological assessment with:
  * NADL-F
  * Frontal Assessment Battery (FAB)
  * functional scales assessing activities of daily living (ADL) and instrumental activities of daily living (I-ADL)
  * Mini-Mental Parkinson (MMP) - For Parkinson's Disease patients
  * Montreal Cognitive Assessment (MoCA) - for brain tumor and stroke patients

SUMMARY:
The present project aims to investigate the financial capacity in patients diagnosed with Parkinson's Disease or parkinsonism, brain tumor (glioma or meningioma) and cerebrovascular lesion (stroke), in order to evaluate the presence and degree of impairment, and the role of some factors as potential predictors of financial incapacity.

The term 'financial capacity' means both operations relating, for example, to asset management or investing money, and activities of daily life such as shopping or using small sums of money; these activities are mediated by different cognitive functions, from numerical and arithmetic skills to decision making. Financial capacity is, in fact, an instrumental activity of daily life (i.e. Instrumental Activity Of Daily Living, I-ADL) whose impairment negatively affects the functional autonomy of the individual, so as to be subject to legal protection.

To assess financial capacity, the Numerical Activities of Daily Living - Financial (NADL-F; Arcara et al., 2017) will be administered, a battery of tests aimed at investigating both financial performance and financial competence according to the most recent neuropsychological models proposed in the literature.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* Clinical diagnosis of interest for clinical groups
* For stroke patients: disease duration > 1 month

Exclusion Criteria:

* Other brain disorders different from those of interest
* Sensory-motor deficits that could prevent neuropsychological assessment
* Language disorders that could prevent neuropsychological assessment
* Global cognitive impairment as indexed by MoCA < 26 or MMP < 22.85

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patients with Parkinson's Disease/parkinsonisms
  * Patients with brain tumor
  * Patients with stroke
  * Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2021-08-04 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Numerical Activity of Daily Living Financial (NADL-F) in Patients with Parkinson's Disease/Parkinsonisms | At baseline
  Assessment of financial capacity; score range=0-62; higher scores indicate higher financial capacities
Numerical Activity of Daily Living Financial (NADL-F) in Patients with ischemic or haemorrhagic stroke | At baseline
  Assessment of financial capacity; score range=0-62; higher scores indicate higher financial capacities
Change from baseline in Numerical Activity of Daily Living - Financial (NADL-F)Patients with brain tumors | At 3 and 12 months follow up
  Assessment of financial capacity; score range=0-62; higher scores indicate higher financial capacities
Montreal Cognitive Assessment (MoCA) | At baseline
  Assessment of global cognitive functioning
Frontal Assessment Battery (FAB) | At baseline
  Assessment of global cognitive functioning
Activities of daily living questionnaire (ADL) | At baseline
  Assessment of function independence in everyday life

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Lombardy, Italy

REFERENCES:
- [Background] Arcara G, Burgio F, Benavides-Varela S, Toffano R, Gindri P, Tonini E, Meneghello F, Semenza C. Numerical Activities of Daily Living - Financial (NADL-F): A tool for the assessment of financial capacities double dagger. Neuropsychol Rehabil. 2019 Aug;29(7):1062-1084. doi: 10.1080/09602011.2017.1359188. Epub 2017 Sep 7. PMID 28880732